CLINICAL TRIAL: NCT03099603
Title: A First in Human, Randomized, Double-Blind Study to Assess Safety, Tolerability, and Pharmacokinetics of Single, Ascending Doses of HTD1801 in Healthy Subjects
Brief Title: A Study of HTD1801 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1801.PCT002
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.5g (Placebo Comparator): single dose of placebo to 2 healthy subjects or 0.5g HTD1801 to 6 healthy subjects
  Interventions: Drug: HTD1801
- 1.0g (Placebo Comparator): single dose of placebo to 2 healthy subjects or 1.0g HTD1801 to 6 healthy subjects
  Interventions: Drug: HTD1801
- 2.0g (Placebo Comparator): single dose of placebo to 2 healthy subjects or 2.0g HTD1801 to 6 healthy subjects
  Interventions: Drug: HTD1801
- 4.0g (Placebo Comparator): single dose of placebo to 2 healthy subjects or 4.0g HTD1801 to 6 healthy subjects
  Interventions: Drug: HTD1801

INTERVENTIONS:
Drug: HTD1801 — A small molecular compound for the treatment of primary sclerosing cholangitis

SUMMARY:
This is a randomized, double blind, single center, ascending single dose study to evaluate the safety, tolerability, and PK of HTD1801.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 to ≤ 50 years
2. Body mass index (BMI) ≥18.0 to ≤ 30.0 kg/m2
3. Current non-user of any nicotine containing products (>6 months)
4. Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or post-menopausal for ≥12 months. The site will try to retrieve medical records to document the sterility, however, the absence of records will not exclude screening the participant. If medical records cannot be obtained, serum and urine pregnancy testing will be conducted. Postmenopausal status will be confirmed through testing of FSH levels ≥ 40 IU/mL at screening for amenorrheic female participants <50 years of age.

   Males must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent or if engaged in sexual relations with a child-bearing potential, the participant and his partner must be using an acceptable, highly effective, contraceptive method from Screening and for a period of 60 days after the last dose of Study Drug. Acceptable methods of contraception are the use of condoms and an effective contraceptive for the female partner that includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, or intrauterine contraception/device). The Principal Investigator will assess the adequacy of methods of contraception on a case-by-case basis.
5. Ability to provide written informed consent.

Exclusion Criteria:

1. Participation in an investigational drug study within 30 days prior to dosing or 5 half-lives within the last dose of investigational product whichever is longer.
2. Current use of any prescription or over-the-counter (OTC) medications, including herbal products and supplements, within 14 days prior to Day 1 or 5 half-lives, whichever is longer. [Use of ≤2 g per day of paracetamol (acetaminophen) is allowed prior to and during the study at Investigator discretion. The reason for use must be listed either in the subject's baseline information or as an adverse event.]
3. Any use of non-steroid anti-inflammatory drugs (NSAIDs) within 7 days prior to dosing.
4. History of any serious adverse reaction or hypersensitivity to any of the product components.
5. Use of parenterally administered proteins or antibodies within 12 weeks of screening. (Note: Influenza vaccine will be allowed)
6. Glucose-6-phosphate dehydrogenase(G6PD) deficiency.
7. History of weight loss > 5% in the 8 weeks prior to screening.
8. History of any active infection, other than mild viral illness, within 30 days prior to dosing.
9. History of alcohol or illicit drug abuse as judged by the Investigator within approximately 1 year
10. Use of any nicotine-containing product within 6 months prior to Screening or at any time during the study and follow-up as confirmed by urine cotinine screening.
11. Presence of clinically significant medical history, physical, laboratory, or ECG findings that, in the opinion of the Investigator, may potentially compromise the safety of the subject, or interfere with any aspect of study conduct or interpretation of results.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) after single dose | up to Day 30
  Incidence, severity and causality of AEs and SAEs

SECONDARY OUTCOMES:
HTD1801 plasma concentration levels after single dose | 96 hours
  Concentration-Time data
Pharmacokinetics (PK) of HTD1801 in plasma after single dose - peak plasma concentration (Cmax) | 96 hours
  PK parameters: Cmax
PK of HTD1801 in plasma after single dose - area under the plasma concentration vs. time curve (AUC) | 96 hours
  PK parameters: AUC
PK of HTD1801 in plasma after single dose - time to peak plasma concentration (Tmax) | 96 hours
  PK parameters: Tmax
PK of HTD1801 in plasma after single dose - half life (T1/2) | 96 hours
  PK parameters: T1/2

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wong, Doctor, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Not provided